CLINICAL TRIAL: NCT01702064
Title: A Phase I Study of Ruxolitinib in Combination With Nilotinib in CML Patients With Evidence of Molecular Disease
Brief Title: Ruxolitinib in Combination With Nilotinib in Chronic Myeloid Leukemia (CML) Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-17114
Record Dates: First submitted 2012-10-03; First posted 2012-10-05 (Estimated); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Chronic Phase Chronic Myeloid Leukemia
Keywords: CML; CP-CML; Chronic Phase-CML (CP-CML); chronic myeloid leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — nilotinib; ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nilotinib with Ruxolitinib (Experimental): The starting dose of ruxolitinib will be 5mg by mouth (PO) twice a day (BID) and will increase by 5 mg increments in each cohort, to a maximum dose of 15 mg PO BID. Nilotinib will be given at a dose ranging from 300 mg PO BID to 400 mg PO BID, depending on the participant's dose prior to enrollment on the trial.
  Dose Level 1: Ruxolitinib 5 mg twice a day (BID); Nilotinib 300 mg or 400 mg BID.
  Dose Level 2: Ruxolitinib 10 mg BID; Nilotinib 300 mg or 400 mg BID.
  Dose Level 3: Ruxolitinib 15 mg BID; Nilotinib 300 mg or 400 mg BID.
  Interventions: Drug: Nilotinib; Drug: Ruxolitinib

INTERVENTIONS:
Drug: Nilotinib — Participants will remain on the same dose of nilotinib they have been receiving prior to enrollment on the trial. This will range from 300 mg PO BID to 400 mg PO BID.
  Dose modifications will not occur, as the purpose of this study is to determine the maximum tolerated dose of ruxolitinib, based on the number of dose.
  Other Names: Tasigna; BCR-ABL kinase inhibitor
Drug: Ruxolitinib — Dose escalation will follow a 3+3 study design. Dose modifications will not occur, as the purpose of this study is to determine the maximum tolerated dose, based on the number of dose limiting toxicities seen at a specific dose.
  Other Names: INCB018424

SUMMARY:
This study is designed to determine the maximal tolerated dose of Ruxolitinib in combination with nilotinib in patients with chronic myeloid leukemia (CML).

ELIGIBILITY:
Inclusion Criteria:

* Must have chronic phase chronic myeloid leukemia (CML). They must also be under treatment with nilotinib as either first, second, or third-line therapy.
* Must have a complete cytogenetic response (CCyR) OR must have been on nilotinib for a minimum of 6 months.
* Must not have undergone treatment for any other form of cancer (aside from non-melanoma skin cancer) in the past 5 years.
* 18 years of age or older and must be able to speak and read English or Spanish.
* Able to provide informed consent.
* Prior therapy with a tyrosine kinase inhibitor (TKI) other than nilotinib is allowable, however, nilotinib must be the current therapy. All participants must be under the care of a Moffitt Cancer Center physician, and enrollment is expected to be complete within 6 months.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2 (Karnofsky ≥60%.
* Must have normal organ and marrow function as defined in study protocol.
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of Ruxolitinib and nilotinib administration. Women of child-bearing age will be required to have a negative pregnancy test within 14 days of enrolling in this study.
* Ability to understand and the willingness to sign a written informed consent document
* B-HCG will be performed on all women of child-bearing potential as screening prior to enrollment on this trial. STAT3 levels in the bone marrow will also be measured prior to enrollment.

Exclusion Criteria:

* Patients who are in accelerated phase or blast phase CML.
* May not be receiving any other investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ruxolitinib or other agents used in the study.
* Known history of a prolonged QT interval (QTc >480).
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study. Women who are breast feeding their infants should discontinue this practice if the mother is treated with ruxolitinib.
* Currently receiving any drugs considered to be strong CYP3A4 inducers or inhibitors which cannot be discontinued or changed to an alternative drug prior to enrolling on the trial.
* HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study.
* Patients receiving nilotinib 200 mg by mouth, twice a day (PO BID) or a lower dose are not eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-02-21 (Actual); Primary Completion 2016-10-17 (Actual); Study Completion 2019-01-09 (Actual)

PRIMARY OUTCOMES:
Phase I: Maximum Tolerated Dose (MTD) | Average of 6 months
  Maximum tolerated dose (MTD) of ruxolitinib with nilotinib. Dose escalation will follow a 3+3 study design. If 2 or more participants within a cohort experience a dose limiting toxicity (DLT), then the MTD will have been exceeded and the preceding dose level will be evaluated as the MTD. A minimum of 6 participants must be evaluated at the dose level in order for it to be declared as the MTD.
  Dose limiting toxicity is defined as:
  * Any non-hematological toxicity ≥ grade three, excluding any untreated nausea, vomiting, diarrhea or fatigue that occurs during the first 56 days of therapy.
  * Grade three thrombocytopenia with active bleeding or grade four thrombocytopenia or febrile neutropenia (ANC <500 cells/µL and fever > 101.0 F (38.5C)).
  * Any treatment related grade five toxicity (i.e., death).

OTHER OUTCOMES:
Complete Molecular Response Rate | Up to 36 months
  Complete molecular response rate (CMR >4.5 log reduction) after the treatment combination.

CONTACTS AND LOCATIONS:
Overall Officials: Kendra Sweet, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- [Derived] Sweet K, Hazlehurst L, Sahakian E, Powers J, Nodzon L, Kayali F, Hyland K, Nelson A, Pinilla-Ibarz J. A phase I clinical trial of ruxolitinib in combination with nilotinib in chronic myeloid leukemia patients with molecular evidence of disease. Leuk Res. 2018 Nov;74:89-96. doi: 10.1016/j.leukres.2018.10.002. Epub 2018 Oct 9. PMID 30340199